CLINICAL TRIAL: NCT00345969
Title: Exercise and Testosterone Therapy in Elderly Men With Physical Frailty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Ellen F. Binder, MD, Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC 02-1108
Record Dates: First submitted 2006-06-27; First posted 2006-06-29 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-01

CONDITIONS: Physical Frailty; Hip Fracture; Elective Hip Replacement; Hypogonadism
Keywords: Testosterone Replacement Therapy; Physical Frailty; Hip Fracture
MeSH Terms: conditions — Hip Fractures; Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transdermal Testosterone gel (1%) (Active Comparator): Transdermal testosterone 1% gel (Androgel) provided as 2.5 gm and/or 5 gm gel packets with dose titration and monthly dose adjustments to achieve and maintain serum total testosterone level between 500-900 mg/dL. Gel to be applied daily by participants. Participants are blinded to the contents of the gel packets. Participants in this arm also perform supervised exercise training for 6 months.
  Interventions: Drug: Transdermal Testosterone gel (1%); Behavioral: Supervised exercise training
- Placebo gel (Placebo Comparator): Inactive topical gel identical in appearance to the active medication, provided in packets identical to the packaging for the active medication. Gel to be applied daily by participants. Participants are blinded to the contents of the gel packets. Participants in this arm also perform supervised exercise training for 6 months.
  Interventions: Behavioral: Supervised exercise training

INTERVENTIONS:
Drug: Transdermal Testosterone gel (1%) — Transdermal testosterone replacement therapy with Androgel(TM). Daily application of gel at 5 mg, 7.5 gm, or 10 gm for six months. Target serum total testosterone level between 500-900 ng/dl.
  Other Names: Androgel
  Arms: Transdermal Testosterone gel (1%)
Behavioral: Supervised exercise training — Supervised exercise training performed on site at academic medical center exercise facility. Exercise training consisted of 2 months of flexibility, balance, treadmill walking, and physical therapy-type exercises, followed by 4 months of progressive resistance training.

SUMMARY:
The primary aim of this study is to determine, in hypogonadal older men with physical frailty, whether exercise training combined with testosterone replacement therapy can improve skeletal muscle strength, and lean mass, to a greater degree than exercise training alone.

DETAILED DESCRIPTION:
Decreases in physical abilities, including losses of strength, endurance, balance, and coordination are major causes of disability and loss of independence in older men. Such individuals are at high risk for injurious falls, hospitalization, and use of supportive services. Age-associated testosterone deficiency may contribute to deficits in muscle mass and strength that are common in this patient population.

The primary aim of this study is to determine, in hypogonadal older men with physical frailty, whether six months of exercise training combined with testosterone replacement therapy can improve skeletal muscle mass and skeletal muscle strength, to a greater degree than six months of exercise training alone.

Secondary study aims are to determine in hypogonadal older men with physical frailty, whether six months of exercise training combined with testosterone replacement therapy can improve physical function, bone mineral density, and quality of life, to a greater degree than six months of exercise training alone.

Comparison: Men age 65 years and older who meet criteria for physical frailty and have a serum testosterone level below 350 ng/dl are randomly assigned to one of two groups: 1) transdermal testosterone replacement therapy + supervised exercise training for six months vs. 2) inactive placebo gel + supervised exercise training for six months.

ELIGIBILITY:
Inclusion Criteria:

* Male, age 65 years and older
* Total serum testosterone level < 350 ng/dl
* Total Modified Physical Performance Test Score <28

Exclusion Criteria:

* Inability to walk 50 feet independently
* Current use of estrogen, progestin, or androgen containing compound
* Diagnosis of dementia of severity sufficient to interfere with informed consent or compliance with the protocol, or a score of 11 or greater on the Short Blessed Test of Orientation, Memory and Concentration
* Visual or hearing impairments that interfere with following directions
* Cardiopulmonary disease (recent MI, unstable angina or CHF, etc.), neuromuscular impairments, or unstable medical condition that would contraindicate progressive resistance exercise training
* History of prostate cancer or hormone dependent neoplasia
* PSA level > 4 ng/ml
* Serum liver transaminase levels of greater than 2 standard deviations above normal
* Use of drugs for osteoporosis for less than 1 year
* Current participation in a vigorous exercise or weight-training program more than once per week
* History of sleep apnea requiring use of CPAP
* Uncontrolled thyroid disease
* Diagnosis of cancer within the past 5 years other than superficial skin cancer (squamous or basal cell)
* hematocrit > 50%
* AUA symptom score > 16.
* History of alcohol or substance abuse
* Presence of severe facial acne
* Active symptoms of depression with GDS score > 5 and symptoms severe enough to cause >5% weight loss in previous 3 months or interfere with research assessments

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-11; Primary Completion 2009-02 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen F. Binder, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from orthopedic units of local hospitals, rehabilitation facilities (both acute rehabilitation units and SNFs), home care programs, and the community-at-large.
Pre-assignment Details: Participants were carefully screened for exclusion criteria prior to randomization.
Groups:
- Exercise + Placebo: Participants assigned to this group were prescribed an inactive topical gel for 6 months, and also performed a supervised exercise training program three times per week for 6 months.
- Exercise + Testosterone: Participants assigned to this group were prescribed transdermal testosterone (Androgel 1%) for six months, and performed a supervised exercise training program three times per week for six months.
Period: Overall Study
Arm/Group | Exercise + Placebo | Exercise + Testosterone
Started | 12 | 13
Completed | 11 | 11
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Population: Men who completed the intervention and provided baseline and follow-up data for primary outcome measures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise + Placebo | Exercise + Testosterone | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 81 (4) | 77 (6) | 80 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 11 | 11 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 11 | 9 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Total Modified Physical Performance (mPPT) score [Mean (Standard Deviation); unit: units on a scale] — Range 0-36, (min-max); higher scores indicate better physical performance. The Total mPPT score is constructed by summing sub-scores of 9 performance tasks. Sub-scores have a range of 0-4 (min-max); higher sub-scores indicate better performance.
  units on a scale | 23 (4) | 26 (3) | 25 (4)
Total Testosterone level (ng/dL) [Mean (Standard Deviation); unit: ng/dL] | 252 (71) | 248 (97) | 250 (84)
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 28 (3) | 29 (5) | 29 (4)
Body Weight (lbs.) [Mean (Standard Deviation); unit: lbs.] | 193 (30) | 195 (38) | 194 (34)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Total Lean Body Mass
Description: Total Lean Mass measured by Dual X-ray Absorptiometry (DXA)
Time Frame: Baseline and Six Months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Exercise + Placebo | Exercise + Testosterone
Number analyzed (Participants) | 11 | 11
kg | 0.5 (1.8) | 2.3 (1.0)
Statistical Analysis 1: Comparison: Exercise + Placebo vs Exercise + Testosterone; Test type: Superiority or Other; p = 0.01, ANOVA

2. Primary Outcome: Change in Skeletal Muscle Strength by 1-RM
Description: One-repetition maximum strength for leg extension
Time Frame: Baseline and Six Months
Population: Only 8 participants in the Exercise+Testosterone group provided Leg Extension 1-RM measurements at baseline and 6-month follow-up.
Measure: Mean (Standard Deviation); unit: lbs.
Arm/Group | Exercise + Placebo | Exercise + Testosterone
Number analyzed (Participants) | 11 | 8
lbs. | 59.2 (33.3) | 70.3 (37.5)
Statistical Analysis 1: Comparison: Exercise + Placebo vs Exercise + Testosterone; Test type: Superiority or Other; p = 0.55, ANOVA

3. Secondary Outcome: Change in Isokinetic Leg Extension Torque at 0 Deg/Sec
Description: Leg Extension Torque measured with Cybex dynamometer at 0 deg/sec
Time Frame: Baseline and Six Months
Population: Only 10 participants in Exercise+Placebo group, and 8 participants in Exercise+Testosterone group, provided Leg Extension torque measurements at baseline and 6-month follow-up.
Measure: Mean (Standard Deviation); unit: ft/lb
Arm/Group | Exercise + Placebo | Exercise + Testosterone
Number analyzed (Participants) | 10 | 8
ft/lb | 10.4 (14.2) | 19.8 (18.1)
Statistical Analysis 1: Comparison: Exercise + Placebo vs Exercise + Testosterone; Test type: Superiority or Other; p = 0.23, ANOVA

4. Secondary Outcome: Change in Leg Extension Torque at 60 Deg/Sec
Description: Leg Extension Torque measured with Cybex dynamometry at 60 deg/sec
Time Frame: Baseline and Six Months
Population: Only 10 participants in the Exercise+Placebo group, and 8 participants in the Exercise+Testosterone group, provided Leg extension torque measurements at baseline and 6 month follow-up.
Measure: Mean (Standard Deviation); unit: ft/lb
Arm/Group | Exercise + Placebo | Exercise + Testosterone
Number analyzed (Participants) | 10 | 8
ft/lb | 12.7 (13.5) | 19.4 (21.4)
Statistical Analysis 1: Comparison: Exercise + Placebo vs Exercise + Testosterone; Test type: Superiority or Other; p = 0.43, ANOVA

5. Secondary Outcome: Change in Total Body Fat Mass
Description: Total Body Fat Mass as measured by DXA
Time Frame: Baseline and Six Months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Exercise + Placebo | Exercise + Testosterone
Number analyzed (Participants) | 11 | 11
kg | -0.51 (0.96) | -1.1 (1.7)
Statistical Analysis 1: Comparison: Exercise + Placebo vs Exercise + Testosterone; Test type: Superiority or Other; p = 0.33, ANOVA

6. Secondary Outcome: Change in Femoral Bone Mineral Density (BMD)
Description: Femoral Bone Mineral Density measured with Dual X-ray Absorptiometry (DXA)
Time Frame: Baseline and Six Months
Population: Only 10 participants in the Exercise+Placebo group, and 10 participants in the Exercise+Testosterone group, provided femoral bone density measurements at baseline and the 6 month follow-up.
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | Exercise + Placebo | Exercise + Testosterone
Number analyzed (Participants) | 10 | 10
g/cm2 | -0.008 (1.238) | 0.084 (3.515)
Statistical Analysis 1: Comparison: Exercise + Placebo vs Exercise + Testosterone; Test type: Superiority or Other; p = 0.93, ANOVA

7. Secondary Outcome: Change in Total Modified Physical Performance (mPPT) Score
Description: The Modified Physical Performance Test (mPPT) is a direct observational test that assesses multiple dimensions of physical function (basic and complex activities of daily living [ADL]) with different levels of difficulty. The test consists of 9 performance tasks. The total score range is 0-36 (min-max), with higher scores indicating better performance. Sub-scores are assigned for each of 9 item tasks; sub-score range is 0-4 (min-max) with higher scores indicating better performance. The sub-scores are summed to compute the total score.
Time Frame: Baseline and Six Months
Population: Only 10 participants in the Exercise+Placebo group, and 9 participants in the Exercise+Testosterone group, provided baseline and follow-up mPPT measurements.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise + Placebo | Exercise + Testosterone
Number analyzed (Participants) | 10 | 9
units on a scale | 5.0 (3.7) | 2.8 (4.4)
Statistical Analysis 1: Comparison: Exercise + Placebo vs Exercise + Testosterone; Test type: Superiority or Other; p = 0.24, ANOVA

8. Other Pre Specified Outcome: Change in Serum Prostate Specific Antigen (PSA) Level
Time Frame: Baseline and Six Months
Population: Only 10 participants in the Exercise+Placebo group, and 9 participants in the Exercise+Testosterone group, provided serum PSA level measurements at baseline and 6 month follow-up.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Exercise + Placebo | Exercise + Testosterone
Number analyzed (Participants) | 10 | 9
ng/mL | 0.05 (0.27) | 0.21 (0.63)
Statistical Analysis 1: Comparison: Exercise + Placebo vs Exercise + Testosterone; Test type: Superiority or Other; p = 0.49, ANOVA

9. Other Pre Specified Outcome: Change in Hematocrit
Description: Percentage of the volume of whole blood composed of Red Blood Cells
Time Frame: Baseline and Six Months
Population: Only 10 participants in the Exercise+Placebo group, and 9 participants in the Exercise+Testosterone group, provided hematocrit measurements at baseline and 6-month follow-up.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Exercise + Placebo | Exercise + Testosterone
Number analyzed (Participants) | 10 | 9
percent | 0.14 (2.6) | 2.5 (4.8)
Statistical Analysis 1: Comparison: Exercise + Placebo vs Exercise + Testosterone; Test type: Superiority or Other; p = 0.19, ANOVA

10. Other Pre Specified Outcome: Change in Serum Total Cholesterol Level
Time Frame: Baseline and Six Months
Population: Only 9 participants in the Exercise+Placebo group, and 9 participants in the Exercise+Testosterone group, provided serum for cholesterol measurements at baseline and 6 months.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exercise + Placebo | Exercise + Testosterone
Number analyzed (Participants) | 9 | 9
mg/dL | -3.2 (15.4) | -9.0 (42.9)
Statistical Analysis 1: Comparison: Exercise + Placebo vs Exercise + Testosterone; Test type: Superiority or Other; p = 0.71, ANOVA

11. Other Pre Specified Outcome: Change in Serum HDL Cholesterol Level
Time Frame: Baseline and Six Months
Population: Only 9 participants in the Exercise+Placebo group, and 9 participants in the Exercise+Testosterone group, provided serum for HDL cholesterol measurements at baseline and 6 months.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exercise + Placebo | Exercise + Testosterone
Number analyzed (Participants) | 9 | 9
mg/dL | -1.4 (9.0) | 1.7 (7.8)
Statistical Analysis 1: Comparison: Exercise + Placebo vs Exercise + Testosterone; Test type: Superiority or Other; p = 0.44, ANOVA

12. Other Pre Specified Outcome: Change in Serum LDL Cholesterol Level
Time Frame: Baseline and Six Months
Population: Only 9 participants in the Exercise+Placebo group, and 9 participants in the Exercise+Testosterone group, provided serum for LDL cholesterol measurements at baseline and 6 months.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exercise + Placebo | Exercise + Testosterone
Number analyzed (Participants) | 9 | 9
mg/dL | -3.6 (15.3) | -1.6 (39.0)
Statistical Analysis 1: Comparison: Exercise + Placebo vs Exercise + Testosterone; Test type: Superiority or Other; p = 0.89, ANOVA

13. Secondary Outcome: Change in Serum Testosterone Level
Description: Total Serum Testosterone Level (ng/mL)
Time Frame: Baseline and Six Months
Population: Only 9 participants in the Exercise+Testosterone group provided serum testosterone levels at baseline and 6-month follow-up.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Exercise + Placebo | Exercise + Testosterone
Number analyzed (Participants) | 11 | 9
ng/mL | -15.3 (72.6) | 121.2 (235.5)
Statistical Analysis 1: Comparison: Exercise + Placebo vs Exercise + Testosterone; Test type: Superiority or Other; p = 0.13, ANOVA

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Exercise + Placebo | Exercise + Testosterone
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/13
Other Adverse Events (participants affected / at risk) | 1/12 | 1/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise + Placebo (N=12) | Exercise + Testosterone (N=13)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) — Participant experienced new onset atrial fibrillation that required acute care hospitalization. The patient's symptoms occurred at rest and were not coincident with performing exercise.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise + Placebo (N=12) | Exercise + Testosterone (N=13)
Elevated serum PSA level (Renal and urinary disorders) | 0 (0) | 1 (1) — Participant had elevated PSA level (7.2 ng/mL) at month 6 of study, which returned to normal at 30-day follow up.
Fall (General disorders) | 1 (1) | 0 (0) — Participant experienced a fall during balance testing; no injury sustained.

LIMITATIONS AND CAVEATS:
Small number of subjects enrolled, single site trial, included both hip fracture patients and a few patients with elective hip joint replacement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less